CLINICAL TRIAL: NCT06497790
Title: German Translation and Validation of the Barnes-Jewish-Hospital Stroke Dysphagia Screen (BJH-SDS)
Brief Title: BJH-SDS Validation of the German Translation
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: BJH-G
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Dysphagia; Stroke, Acute
Keywords: Stroke; Dysphagia; Swallowing disorders; FEES; Swallow screening
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute stroke patients: All patients of the participating clinics who have a suspected diagnosis of stroke
  Interventions: Diagnostic Test: BJH-SDS Screenint Test; Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing
- Non-neurologic ICU patients: All patients of the participating clinics who are being treated in intensive care due to a non-neurological disease
  Interventions: Diagnostic Test: BJH-SDS Screenint Test; Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing
- Non-neurologic patientes: All patients of the participating clinics who are being treated due to a non-neurological disease
  Interventions: Diagnostic Test: BJH-SDS Screenint Test; Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Diagnostic Test: BJH-SDS Screenint Test — The test includes the assessment of a sufficient level of consciousness (Glasgow Coma Scale over 13 points), a check for facial paresis, soft palate paresis and tongue paresis followed by a water swallow test with 90 ml of water if the previous points are assessed as normal. The water swallow test checks for signs of aspiration (throat clearing, coughing or a change in voice quality)
Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing — The FEES evaluates anatomical changes, functional disorders of the visible structures (e.g. recurrent paresis), saliva management, penetration and aspiration of food boluses in order to draw conclusions about the underlying pathomechanism of dysphagia. It is an established standard diagnostic procedure for stroke patients and, in addition to the diagnosis of dysphagia, also enables pathomechanism-guided therapy by speech therapists
  Other Names: FEES

SUMMARY:
The first object of the study is the validation of a translation of the Barnes-Jewish Hospital Stroke Dysphagia Screen with determination of sensitivity, specificity, interrater reliability (especially between different professional groups) and criterion validity.

If the German translation proves to be suitable, it will also be validated on general neurological patients, i.e. patients on a neurological ward without a stroke.

DETAILED DESCRIPTION:
Stroke is now the second most common cause of death worldwide. Dysphagia is described as a direct consequence of cerebral infarction in at least 50% of stroke patients in the acute phase [2]. It often leads to aspiration pneumonia, which is the most important secondary complication in stroke unit. Within one year after a stroke, around 20% of dysphagia patients die as a result of aspiration pneumonia . In addition, dysphagia causes numerous other secondary complications (malnutrition, exsiccosis) and associated high costs for the healthcare system.

Numerous screening procedures have been developed in recent years. These are mostly based on a swallowing test with water after testing various input requirements. There are also multi-consistency tests that include liquids as well as pulpy and solid consistencies. The sensitivity of the tests is usually at least 85% with moderate specificity, which is due to the inability to detect silent aspiration by non-instrumental diagnostics. In addition, the implementation of the screening procedures is usually only evaluated by the professional group of speech therapists.

One of these screening procedures is the Barnes-Jewish-Hospital Stroke Dysphagia Screen (BJH-SDS). In our opinion, this test is very well suited as a screening procedure, as it has good sensitivity (94%) and specificity (64%), is validated for all professional groups and takes little time. In brief, it includes an assessment of sufficient consciousness (Glasgow Coma Scale over 13 points), a check for facial paresis, soft palate paresis and tongue paresis followed by a water swallow test with 90 ml of water if the previous points are assessed as normal. The water swallow test checks for signs of aspiration (throat clearing, coughing or a change in voice quality) However, the BJH-SDS is not yet available in German. The aim of this research project is therefore to translate the BJH-SDS into German (BJH-SDS-G) and validate it as the gold standard using flexible endoscopic swallowing examination (FEES) and then use it routinely in our clinics. This will be followed by validation in general neurological patients (without stroke) so that the BJH-SDS can also be used reliably in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* All stroke patients in the neurology department of the Lahn-Dill Clinic in Wetzlar and the stroke unit of the Bürgerhospital in Friedberg and the neurologic ICU of the University Hospital in Giessen are to be screened with the BJH-SDS-G after appropriate information has been provided.

Exclusion Criteria:

* Exclusion criteria are a lack of informed consent, contraindications to an FEES examination, a history of stroke, pre-existing dysphagia or a disease that may be associated with dysphagia (e.g. ENT tumors, Parkinson's disease, neuromuscular diseases).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Acute ischemic stroke Patients
  * General patient popluation
  * Non-neurologic ICU patients
Sampling Method: Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Score | Immediately after the intervention
  Penetration-Aspiration-Score, minimum value 1, maximum value 8; higher scores mean worse outcome
Barthel-Index | Immediately before the intervention
  Barthel-Index; minimal value 0, maximum value 100; lower values mean worse outcome
MRS | Immediately before the intervention
  Modified Rankin Scale; minimal value 0, maximum value 6; higher values mean worse score

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Braun, PD MD, Study Director — University of Giessen; Samra Hamzic, Dr., Principal Investigator — University of Giessen
Locations (1):
- University Hospital Giessen and Marburg, Campus Giessen, Giesen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided